CLINICAL TRIAL: NCT05009199
Title: A Phase 1 Proof of Principle Study to Evaluate the Occupancy of A2A Receptors Using PET Radiotracer [18F]MNI-444 & Repeated Dosing of Oral Caffeine in Participants Without Parkinson's Disease Who Carry Pathogenic Mutation in the LRRK2 Gene
Brief Title: Occupancy of Adenosine A2A Receptors Using the PET Radiotracer [18F]MNI-444
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Invicro (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: [18F]MNI-444 (9564)
Record Dates: First submitted 2021-07-01; First posted 2021-08-17 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-07

CONDITIONS: Healthy Volunteer
Keywords: HV
MeSH Terms: interventions — MNI-444

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]MNI-444 (Experimental): After a wash-out of caffeine of at least 24 hours, each participant will receive a single injection of [18F]MNI-444 followed by brain PET imaging of up to 90 minutes to establish baseline A2A receptor binding.
  Interventions: Drug: [18F]MNI-444

INTERVENTIONS:
Drug: [18F]MNI-444 — Subjects will undergo PET imaging using [18F]MNI-444.

SUMMARY:
The overall goal of this protocol is to evaluate the binding of caffeine to adenosine A2A receptors in the brain of participants at risk for developing PD.

DETAILED DESCRIPTION:
The overall goal of this protocol is to evaluate the binding of caffeine to adenosine A2A receptors in the brain of participants at risk for developing PD. The specific objectives are:

* To evaluate the pharmacokinetics (PK) and pharmacodynamics of multiple doses of oral caffeine on striatal binding of the adenosine A2A receptor ligand [18F]MNI-444.
* To evaluate the safety and tolerability of 3 doses of the positron emission tomography (PET) radiotracer, [18F]MNI-444.
* To evaluate the safety and tolerability of multiple doses of oral caffeine in this paradigm.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible for inclusion in this study only if they meet all of the following criteria:

* Participant is able to provide written informed consent, which must be obtained before any assessment is performed.
* Female participants must not be of childbearing potential, or if they are of childbearing potential, must agree to use contraception and not donate eggs. At the discretion of the Investigator, participants without documentation of non-childbearing potential may receive pregnancy testing.

  * A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (ie, removal of ovaries, fallopian tubes, and/or uterus, tubal ligation) or another cause as determined by the Investigator (eg, Müllerian agenesis).
  * Women of childbearing potential must commit to remain abstinent (refrain from heterosexual intercourse) or use 2 forms of birth control, 1 of which is a barrier contraception method, for the duration of the study and 30 days after study completion. Periodic abstinence (eg, calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception.
  * Women of childbearing potential must commit to not donate ovum for the duration of the study and 30 days after study completion.
* Male participants with partners of childbearing potential must commit to the use of 2 methods of contraception, 1 of which is a barrier method for male participants for the study duration and 90 days after study completion.
* Male participants must not donate sperm for the study duration and for 90 days after study completion.
* Willing and able to cooperate with study procedures.
* Males and females aged ≥ 30 years.
* Healthy with no clinically relevant finding on physical examination at Screening.
* No personal history of clinically significant neurologic and/or psychiatric disorders, including PD.
* No history of dopamine transporter deficit on DaTscan for any previously acquired DaTscan.
* No cognitive impairment as judged by the Investigator.
* Has a sequence variation in the LRKK2 gene that is a genetic risk factor for the development of PD (based on previous genetic testing in medical history).

Exclusion Criteria:

Participants fulfilling any of the following criteria are not eligible for inclusion in this study:

* Current or prior history of any alcohol or drug abuse in the past 2 years.
* Laboratory tests with clinically significant abnormalities and/or clinically significant unstable medical illness.
* Participant has received an investigational drug within 30 days or five half-lives prior to the baseline assessments, whichever is longer.
* Prior participation in other research protocols or clinical care during the past year that would result in radiation exposure to an effective radiation dose exceeding the acceptable annual limit established by the US Federal Guidelines (effective dose of 50 mSv, including the procedures in this clinical protocol).
* Pregnant, lactating or breastfeeding.
* Evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Unsuitable veins for repeated venipuncture.
* Brain MRI with clinically significant structural abnormalities.
* Has a medical condition or takes a medication likely to interfere with assessment of brain A2A receptor levels by PET in the opinion of the Investigator.
* Implants such as implanted cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, CNS aneurysm clips and other medical implants that have not been certified for MRI, or history of claustrophobia in MRI, unless a previous MRI is used.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacodynamics of multiple doses of oral caffeine on striatal binding of the adenosine A2A receptor ligand [18F]MNI-444. | 1 year
  A2A receptor occupancy will be assessed by comparing the binding potential (BPND) of [18F]MNI-444 in striatal regions of interest (ROIs) for each post-dose scan (ie, peak and trough scans assessed separately) with the baseline scan in the same participant.
To evaluate the pharmacokinetics of multiple doses of oral caffeine on striatal binding of the adenosine A2A receptor ligand [18F]MNI-444. | 1 year
  Plasma PK samples for caffeine and metabolite paraxanthine will be collected during [18F]MNI-444 PET imaging sessions. These concentrations will be used to help understand the A2A receptor occupancy values.

CONTACTS AND LOCATIONS:
Overall Officials: David Russell, M.D., Ph.D, Principal Investigator — Invicro
Locations (1):
- Invicro, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Information — http://invicro.com